CLINICAL TRIAL: NCT06616233
Title: Effects of Chronic Remote Ischaemic Conditioning on Coronary and Peripheral Vascular Function in Patients With Heart Failure
Brief Title: Remote Ischaemic Conditioning (RIC) in Heart Failure
Acronym: ENRICH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0912
Record Dates: First submitted 2023-11-30; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Type 2 Diabetes; Dilated Cardiomyopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiomyopathy, Dilated | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Randomised trial of the effect of remote ischemic conditioning with or without lower intensity exercise on hyperaemic myocardial blood flow in patients with or at risk of heart failure.
Masking Description: Blinded analysis of data
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischaemic Conditioning with Exercise (Experimental): Participants will be randomised to receive remote ischaemic conditioning (RIC) with exercise involving a 4-week home-based programme of RIC with exercise . The exercise will involve handgrip exercise during the cuff deflation phase of RIC.
  Interventions: Device: Remote Ischaemic Conditioning with exercise
- Remote Ischaemic Conditioning (Other): Participants will receive remote ischaemic conditioning (RIC) without exercise involving a 4-week home-based programme of RIC.
  Interventions: Device: Other: Remote Ischaemic Conditioning

INTERVENTIONS:
Device: Remote Ischaemic Conditioning with exercise — Participants will receive RIC through an automated device that will provide cycles on ischaemia/reperfusion to the target organ (arm). During the cuff deflation phase, participants will undergo handgrip exercise at 20-30% of their maximal voluntary contraction for 3 minutes. There will be a total of 4 cycles of exercise.
  Arms: Remote Ischaemic Conditioning with Exercise
Device: Other: Remote Ischaemic Conditioning — Participants will receive RIC through an automated device that will provide cycles on ischaemia/reperfusion to the target organ (arm).. There will be a total of 4 cycles.
  Arms: Remote Ischaemic Conditioning

SUMMARY:
This study will test the impact of remote ischaemic conditioning combined with exercise on myocardial perfusion in patients with or at risk of heart failure

DETAILED DESCRIPTION:
Heart failure (HF) is a disease which affects the heart's ability to pump or fill with blood. It can affect a person's quality of life and their ability to exercise. Recent work has shown that a reduction in the blood supply to the heart may contribute to the problem. It is therefore possible that improving the blood supply to the heart may help patients with HF. One possible way that this might be achieved is with a method called remote ischaemic conditioning (RIC). This involves placing a cuff on a person's arm (identical to a blood pressure cuff) and inflating it for a few minutes to reduce the blood flow in a person's arm. This is thought to release chemicals into the bloodstream which can have positive effects on the heart. This has been studied in patients with other forms of heart disease, but is yet to be tested properly in patients with heart failure. It is hypothesized that combining the RIC procedure with a low level of arm exercise may result in further improvements in the person's blood vessels and heart. This will be tested in a single-centre prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ability to provide written consent
* clinical diagnosis of HFpEF (LVEF ≥50%; symptoms and signs of heart failure [HF] caused by a structural and/or functional abnormality, and at least one: elevated natriuretic peptides; ambulatory; BNP ≥35 pg/mL or NT-proBNP ≥125 pg/mL or hospitalised; BNP ≥100 pg/mL or NT-proBNP ≥300 pg/mL, and objective evidence of cardiogenic pulmonary or systemic congestion) OR stable type 2 diabetes (determined by formal diagnosis in hospital or GP case records with diagnostic oral glucose tolerance test or glycated haemoglobin level ≥6.5%) and with ACC/AHA stage B HF (structural disorder of the heart but no current or previous symptoms of HF) OR confirmed diagnosis of dilated cardiomyopathy

Exclusion Criteria:

* Absolute contraindications to MRI or contrast (e.g. severe claustrophobia, pregnancy, ferromagnetic implants, inability to lie flat, severe renal impairment eGFR<30ml/min/m2)
* Moderate to severe valvular heart disease
* Confirmed coronary artery disease (>50% narrowing in any major epicardial coronary artery on invasive or computed tomography coronary angiography, previous myocardial infarction, previous percutaneous intervention or coronary bypass surgery)
* Known arterial stenosis of the upper extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Myocardial perfusion reserve | 4 weeks
  myocardial perfusion reserve under adenosine stress as assessed by quantitative cardiovascular magnetic resonance (CMR)
Contraction strength in the cuff deflation phase of RIC | 1 day
  contraction force achieved during cuff deflation phase, measured in Newtons
Hyperaemic myocardial blood flow | 4 weeks
  myocardial blood flow under adenosine stress as assessed by quantitative cardiovascular magnetic resonance (CMR)

SECONDARY OUTCOMES:
Brachial artery flow mediated dilation | 4 weeks
  endothelial function as assessed by vascular ultrasound
Skeletal muscle strength | 4 weeks
  maximal handgrip strength (newtons)
Skeletal muscle endurance | 4 weeks
  Isometric skeletal muscle endurance test assessed using handgrip dynamometer (sec)
Cardiopulmonary exercise test | 4 weeks
  VO2 max for maximal aerobic capacity
Brachial artery maximal dilatory capacity | 4 weeks
  endothelial function in response to Glyceryl trinitrate (GTN) as assessed by vascular ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jayanth R Arnold, BMBCh DPhil, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leics, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD